CLINICAL TRIAL: NCT05793983
Title: The Interaction of the S100A8/A9 Protein With the Innate Immune System in the Immunopathology of Acute and Chronic Liver Disease
Brief Title: S100A8/A9 and Innate Immunity in Liver Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St George's, University of London (Other)
Collaborators: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 2021.0073; 285573 (Other: Integrated Research Application System)
Record Dates: First submitted 2021-10-08; First posted 2023-03-31 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Cirrhosis, Liver; Immune Suppression; Liver Failure, Acute on Chronic; Ascites Hepatic; Infections
Keywords: cirrhosis; acute-on-chronic liver failure; immune paralysis
MeSH Terms: conditions — Liver Cirrhosis; Acute-On-Chronic Liver Failure; Infections; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood including derives peripheral blood mononuclear cells, plasma and serum Ascites and ascitic cells Faecal material Urine Broncho-alveolar lavage fluid Liver tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (11):
- Patients with acute or chronic liver disease: 1. Presence of chronic liver disease, or cirrhosis due to any aetiology (latter based upon a histopathological diagnosis or compatible laboratory data and radiological findings)
  2. Acute alcoholic hepatitis
  3. Acute liver failure due to any aetiology
  4. Acute-on-chronic liver failure
- Patients undergoing diagnostic or therapeutic abdominal paracentesis: Patients with acute or chronic liver disease of any aetiology undergoing clinically-indicated paracentesis for ascites
- Patients undergoing broncho-alveolar lavage: 1. Intubated patients with liver disease in intensive care
  2. Undergoing a bronchoscopy or a non-directed broncho-alveolar lavage as part of their routine clinical care
- Patients with acute or chronic liver disease undergoing liver biopsy
- Patients with undergoing transjugular intrahepatic shunt (TIPSS) placement
- Patients with acute or chronic liver disease undergoing orthoptic liver transplantation
- Patients undergoing surgical liver resection or hepatectomy for liver-related diseases
- Patients with ascites without chronic liver disease: 1. Absence of cirrhosis based on clinical, radiological or histopathological features, including patients with non-cirrhotic portal hypertension, cardiac ascites (ascites due to heart failure) or patients with chronic kidney disease undergoing continuous ambulatory peritoneal dialysis (CAPD)
  2. Presence of clinically significant ascites
  3. Undergoing diagnostic or therapeutic paracentesis
- Patients with sepsis without acute or chronic liver disease
- Patients with haemochromatosis who undergo regular venesection
- Healthy subjects

SUMMARY:
This observational study evaluates the concentration of immune protein S100A8/A9 in different liver failure syndromes, its interaction with the immune system and validity as an immunotherapeutic target to improve survival in patients with advanced cirrhosis and/or acute on chronic liver failure.

DETAILED DESCRIPTION:
A paradox exists in chronic liver disease whereby there is a general recognition that chronic inflammation is part of the pathophysiology, heightened when there is an acute deterioration and organ failure (acute-on-chronic liver failure), yet there is an increased susceptibility to infection due to a dysfunctional immune system, which is often the trigger for organ failure and the reason for death in these patients.

A danger signal reported in other inflammatory conditions called S100A8/A9 (calprotectin) is known to activate the immune system by production of pro-inflammatory cytokines but has also been observed to promote the development immunosuppressive signals (e.g. IL-10 and MDSCs).

In an attempt to explain this paradox in liver disease, this study proposes to identify at the cellular and molecular level, the triggers for S100A8/A9 production, how it varies with time in stable patients and those that have acute deteriorations including the development of organ failure, and its interaction with innate immune cells in the circulation and at tissue level.

By studying this, the Investigators hope to be able to identify immunotherapeutic targets and understand whether potential immunotherapy could be applied locally or systemically. The Investigators' observations in this study could provide the basis for the future development of clinical immunomodulating agents, which may ameliorate immunopathology, reduce susceptibility to infection and could reduce mortality in critically ill patients with liver disease. Findings in this study may also have more generalizable impact especially with the recent recognition in the COVID-19 pandemic that immunomodulatory therapies may improve the clinical outcomes of inflammatory phenotypes in virus-induced severe sepsis.

ELIGIBILITY:
Inclusion Criteria:

A) Patients with acute or chronic liver disease:

1. Presence of chronic liver disease, or cirrhosis due to any aetiology (latter based upon a histopathological diagnosis or compatible laboratory data and radiological findings)
2. Acute alcoholic hepatitis (definition as per Crabb et al, 2016)35
3. Acute liver failure due to any aetiology
4. Acute-on-chronic liver failure (defined as per EASL-CLIF definition)17

B) Patients undergoing diagnostic or therapeutic abdominal paracentesis Patients with acute or chronic liver disease of any aetiology undergoing clinically-indicated paracentesis for ascites

C) Patients undergoing broncho-alveolar lavage

1. Intubated patients with liver disease in intensive care
2. Undergoing a bronchoscopy or a non-directed broncho-alveolar lavage as part of their routine clinical care

D) Patients with acute or chronic liver disease undergoing liver biopsy (percutaneous or transjugular) as routine part of their clinical care

E) Patients with portal hypertension (cirrhotic or non-cirrhotic) undergoing transjugular intrahepatic shunt (TIPSS) placement as part of their routine care

F) Patients with acute or chronic liver disease undergoing orthoptic liver transplantation

G) Patients undergoing surgical liver resection or hepatectomy for liver-related diseases

Control groups:

A) Patients with ascites without chronic liver disease:

1. Absence of cirrhosis based on clinical, radiological or histopathological features, including patients with non-cirrhotic portal hypertension, cardiac ascites (ascites due to heart failure) or patients with chronic kidney disease undergoing continuous ambulatory peritoneal dialysis (CAPD)
2. Presence of clinically significant ascites
3. Undergoing diagnostic or therapeutic paracentesis

B) Patients with sepsis without acute or chronic liver disease

C) Patients with haemochromatosis without liver disease or end-organ damage who undergo regular venesection

D) Healthy subjects

Exclusion Criteria:

Age under 18 or over 80 Evidence of disseminated malignancy (isolated cancers including hepatocellular carcinoma are not an exclusion criteria) Patients with known immunodeficiency syndromes (e.g. HIV infection)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary population is patients with acute or chronic liver disease admitted to hospital (including intensive care unit) or out-patient setting. Control subjects includes patients with sepsis, patients without liver disease but on continuous ambulatory peritoneal dialysis for renal replacement therapy (ascites control) and healthy subjects.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2023-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Concentration of plasma S100A8/A9 | 1 years
  The study will evaluate whether S100A8/A9 concentration can be used to predict clinical outcomes, such as mortality, the development of infection and/or organ failure. In the laboratory, it will evaluate the effect S100A8/A9 has on immune functional readouts including phagocytosis, oxidative burst and cytokine production, all of which are required for an effect immune response. Similarly, by blocking its action, the study will identify whether this is a potential immunotherapeutic strategy to improve the outcome of patients with high concentrations of the protein.

SECONDARY OUTCOMES:
Mortality | 1 years
  28-, 90-day and 1 year mortality and its relationship to baseline and serial S100A8/A9 concentration
Development of infection | 1 years
  Incidence of infection in patients with liver disease and its relationship to baseline or dynamic S100A8/A9 concentration

CONTACTS AND LOCATIONS:
Overall Officials: Arjuna Singanayagam, MBBS; PhD, Principal Investigator — St George's, University of London
Locations (1):
- Arjuna Singanayagam, Wandsworth, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No